CLINICAL TRIAL: NCT02396134
Title: A Phase II Randomized, Placebo-Controlled, Multicenter Trial to Evaluate Protective Function of an Optimized Dose of CMVPepVax in Recipients of an Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: Vaccine Therapy in Reducing the Frequency of Cytomegalovirus Events in Patients With Hematologic Malignancies Undergoing Donor Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 13494; NCI-2015-00283 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13494 (Other: City of Hope Medical Center); R01CA181045 (NIH)
Record Dates: First submitted 2015-03-12; First posted 2015-03-24 (Estimated); Results first posted 2023-07-12 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Hodgkin Lymphoma; Adult Non-Hodgkin Lymphoma; Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Cytomegaloviral Infection; Hematopoietic and Lymphoid Cell Neoplasm; HLA-A*0201 Positive Cells Present; Myelodysplastic Syndrome; Adult Lymphoblastic Lymphoma; Chronic Lymphocytic Leukemia; Myelofibrosis; Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Hodgkin Disease; Lymphoma, Non-Hodgkin; Leukemia, Myeloid, Chronic-Phase; Cytomegalovirus Infections; Hematologic Neoplasms; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Primary Myelofibrosis; Myeloproliferative Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (CMVpp65-A*0201 peptide vaccine) (Experimental): Patients receive CMVpp65-A*0201 peptide vaccine SC on days 28 and 56 after HCT.
  Interventions: Biological: CMVpp65-A*0201 peptide vaccine; Other: Laboratory Biomarker Analysis
- Arm II (placebo) (Placebo Comparator): Patients receive placebo SC on days 28 and 56 after HCT.
  Interventions: Other: Placebo; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: CMVpp65-A*0201 peptide vaccine — Given SC
  Arms: Arm I (CMVpp65-A*0201 peptide vaccine)
Other: Placebo — Given SC
  Other Names: placebo, Placebo, placebo therapy, PLCB, sham therapy
  Arms: Arm II (placebo)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well vaccine therapy works in reducing the frequency of cytomegalovirus severe infections (events) in patients with hematologic malignancies undergoing donor stem cell transplant. Vaccines made from a peptide may help the body build an effective immune response and may reduce cytomegalovirus events after donor stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if cytomegalovirus (CMV) peptide(Pep)vaccine(Vax) (CMVpp65-A*0201 peptide vaccine) increases levels, function and kinetics of CMV-specific T cell immunity in vaccinated compared to placebo treated human leukocyte antigen (HLA) A*0201 allogeneic CMV positive hematopoietic stem cell transplant (HCT) recipients (HCT-R+). (Entire cohort) II. To provide a preliminary evaluation of the incidence of CMV reactivation between day 56 and day 180 in patients who receive standard letermovir (Prevymis) prophylaxis (from day 14 through day 100), comparable to the evaluation of an expansion cohort in a pilot study, or the futility stage of a phase II trial. (Letermovir combination cohort) III. To determine if CMVPepVax increases levels, function and kinetics of CMV-specific T cell immunity in vaccinated HCT patients who receive standard Prevymis prophylaxis. (Letermovir combination cohort)

SECONDARY OBJECTIVES:

I. To determine, within the constraints of a pilot cohort, if CMVPepVax reduces the frequency of CMV events alone or in combination with Prevymis defined as reactivation or CMV disease in HLA A*0201 allogeneic HCT-R+.

II. To evaluate the safety and tolerability of CMVPepVax by assessing the following: non-relapse mortality (NRM) at 100 days post HCT, severe (grade 3-4) acute graft versus host disease (GVHD) (aGVHD), and grade 3-4 adverse events (AEs) (Common Terminology Criteria for Adverse Events [CTCAE] 4.0) probably or definitely related to the vaccination within 2 weeks from each vaccination.

III. To characterize CMV reactivation and CMV disease in recipients of CMVPepVax compared to placebo by assessing time-to viremia (defined as number of days from transplantation to the date of >= 500 CMV gc/mL), duration of viremia, recurrence of viremia, incidence of late CMV viremia/disease (> 100 and =< 360 days post HCT), use of antiviral drugs (triggered by clinically significant viremia), cumulative number of CMV specific antiviral treatment days.

IV. To determine whether vaccination induces adaptive natural killer (NK) cell population changes, and increase in the highly cytotoxic memory NKG2C+ NK cells.

V. To determine the impact of CMVPepVax on CMV immune reconstitution in patients who undergo treatment with antiviral agent Prevymis.

VI. To explore GVHD biomarkers and compare between the vaccine and placebo groups.

VII. To characterize CMV reactivation after day 180

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive CMVpp65-A*0201 peptide vaccine subcutaneously (SC) on days 28 and 56 after HCT.

ARM II: Patients receive placebo SC on days 28 and 56 after HCT.

After completion of study treatment, patients are followed up to day 365 after HCT.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Participant must be willing to comply with study and/or follow-up procedures, including willingness to be followed for one year post-HCT
* Planned HCT for the treatment of the following hematologic malignancies:

  * Lymphoma (Hodgkin and non-Hodgkin)
  * Myelodysplastic syndrome
  * Acute lymphoblastic leukemia in first or second remission (for acute lymphoblastic leukemia/lymphoblastic lymphoma, the disease status needs to be in hematologic remission by bone marrow and peripheral blood; persistent lymphadenopathy on computed tomography [CT] or CT/positron emission tomography [PET] scan without progression is allowed)
  * Acute myeloid leukemia in first or second remission
  * Chronic myelogenous leukemia in first chronic or accelerated phase, or in second chronic phase
  * Other hematologic malignancies including chronic lymphocytic leukemia, myeloproliferative disorders and myelofibrosis; patients with multiple myeloma and those with non-malignant disease such as aplastic anemia are excluded
* HLA A*0201 High resolution, 4-digit typing is required at HLA-A2 to ensure A*0201 status.
* CMV seropositive (recipient)
* Planned related or unrelated HCT, with HLA donor allele matching; related donor must be an 8/8 match for HLA-A, -B, and -C at intermediate (or higher) resolution, and -DRB1 at high resolution using deoxyribonucleic acid (DNA)-based typing; unrelated donor must be an 8/8 match at HLA-A, -B, -C, and -DRB1 at high resolution using DNA-based typing; patients undergoing a second allo HCT are not eligible (patients who have undergone a previous autologous HCT are eligible)
* Planned HCT with no ex-vivo T cell depletion of graft; conditioning and immunosuppressive regimens according to institutional guidelines are permitted
* Negative serum or urine beta-human chorionic gonadotropin (HCG) test (female patient of childbearing potential only) within two weeks of registration
* Seronegative for human immunodeficiency virus (HIV), hepatitis C virus (HCV) and active hepatitis B virus (HBV) (surface antigen negative) within 2 months of registration
* Agreement by females of childbearing potential and sexually active males to use an effective method of contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for up to 90 days post-HCT; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately

Exclusion Criteria:

* Any prior investigational CMV vaccine
* Experimental anti-CMV chemotherapy in the last 6 months
* Planned medications from the time of HCT to day 70 post-HCT:

  * Live attenuated vaccines
  * Medically indicated subunit (Engerix-B for HBV; Gardasil for human papilloma virus [HPV]) or killed vaccines (e.g. influenza, pneumococcal, or allergy treatment with antigen injections)
  * Allergy treatment with antigens injections
  * Alemtuzumab or any equivalent in vivo T-cell depleting agent; this includes anti-thymocyte globulin (ATG) and post-transplant cyclophosphamide
  * Antiviral medications with known therapeutic effects against CMV such as ganciclovir (GCV)/valine (VAL), foscarnet (FOS), cidofovir, hexadecyloxypropyl-cidofovir (CMX-001) and maribavir; acyclovir has no therapeutic efficacy against CMV and is allowable as standard of care to prevent herpes simplex virus (HSV)
  * Other investigational product - concurrent enrollment in other clinical trials using an investigational product is prohibited
  * Other medications that might interfere with the evaluation of the investigational product
* Patients with active autoimmune conditions requiring systemic immunosuppressive therapy within the previous 5 years are not eligible
* Pregnant women and women who are lactating; breastfeeding should be discontinued if the mother is enrolled on this study
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., social/psychological issues, etc
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2018-03-04 (Actual); Study Completion 2024-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryotaro Nakamura, MD, Principal Investigator — City of Hope Medical Center
Locations (5):
- United States (5):
  - City of Hope Medical Center, Duarte, California
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Result] Gooley TA, Leisenring W, Crowley J, Storer BE. Estimation of failure probabilities in the presence of competing risks: new representations of old estimators. Stat Med. 1999 Mar 30;18(6):695-706. doi: 10.1002/(sici)1097-0258(19990330)18:63.0.co;2-o. PMID 10204198

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (CMVpp65-A*0201 Peptide Vaccine) | Arm II (Placebo)
Started | 32 | 29
Completed | 32 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (CMVpp65-A*0201 Peptide Vaccine) | Arm II (Placebo) | Total
Number analyzed (Participants) | 32 | 29 | 61
Age, Continuous [Median (Full Range); unit: years] | 61 [25 to 72] | 64 [28 to 74] | 62 [25 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 5 | 18
  Male | 19 | 24 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 20 | 41
  Hispanic | 9 | 8 | 17
  Asian | 1 | 0 | 1
  Black | 0 | 1 | 1
  Non-disclosed | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 32 | 29 | 61

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of CMV at 100 Days
Description: The primary endpoint was CMV event. A CMV event encompasses detection of CMV by either qPCR (termed "reactivation": DNAemia at ≥500 gc/ml = 1250iu/ml) or by tissue histology (end-organ disease). The cumulative incidence was calculated as competing risks using the method of Gooley with death viewed as a competing risk.
Time Frame: Up to day 100 after HCT
Measure: Number (95% Confidence Interval); unit: cases per 100 persons
Arm/Group | Arm I (CMVpp65-A*0201 Peptide Vaccine) | Arm II (Placebo)
Number analyzed (Participants) | 32 | 29
cases per 100 persons | 25.1 [11.6 to 41.2] | 13.8 [4.2 to 28.9]

2. Secondary Outcome: Non-Relapse Mortality (NRM) at 100 Days
Description: NRM was defined as death without recurrent or progressive disease after transplant. Probabilities of NRM were calculated as competing risks using the method of Gooley with relapse viewed as a competing risk.
Time Frame: Up to 100 days after transplant
Measure: Number (95% Confidence Interval); unit: cases per 100 persons
Arm/Group | Arm I (CMVpp65-A*0201 Peptide Vaccine) | Arm II (Placebo)
Number analyzed (Participants) | 32 | 29
cases per 100 persons | 3.1 [0.2 to 14.0] | 3.4 [0.2 to 15.3]

3. Secondary Outcome: Cumulative Incidence of Relapse at One Year
Description: Probabilities of relapse were calculated as competing risks using the method of Gooley with death viewed as a competing risk.
Time Frame: Up to 365 days after HCT
Measure: Number (95% Confidence Interval); unit: cases per 100 persons
Arm/Group | Arm I (CMVpp65-A*0201 Peptide Vaccine) | Arm II (Placebo)
Number analyzed (Participants) | 32 | 29
cases per 100 persons | 12.5 [3.9 to 26.5] | 25.7 [11.1 to 43.3]

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed up to 100 days post-transplant. All-Cause Mortality monitored/assessed up to 1 year post-transplant.
Arm/Group | Arm I (CMVpp65-A*0201 Peptide Vaccine) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 8/32 | 4/29
Serious Adverse Events (participants affected / at risk) | 10/32 | 7/29
Other Adverse Events (participants affected / at risk) | 28/32 | 26/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (CMVpp65-A*0201 Peptide Vaccine) (N=32) | Arm II (Placebo) (N=29)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 3 (3) | 2 (2)
Hospitalization for worsening GVHD symptoms (General disorders) | 0 (0) | 1 (1)
CMV viremia (Infections and infestations) | 1 (2) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
negative rod bacteremia (Infections and infestations) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 1 (3) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte derangements (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
syncope (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (2) | 0 (0)
Hemorrhagic cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
parainfluenza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Worsening skin GVHD (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (CMVpp65-A*0201 Peptide Vaccine) (N=32) | Arm II (Placebo) (N=29)
Anemia (Blood and lymphatic system disorders) | 21 (91) | 22 (94)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
progression to AML (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
heart palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 2 (2)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (14) | 6 (8)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (2) | 2 (4)
CMV gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (5) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 15 (27) | 12 (21)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (3)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (3) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth lesion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth lesion/sore (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (2)
Nausea (Gastrointestinal disorders) | 16 (33) | 11 (25)
Oral pain (Gastrointestinal disorders) | 1 (1) | 4 (4)
Pearly Papule on oral mucosa (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 8 (9) | 5 (5)
mouth pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
mouth sores (Gastrointestinal disorders) | 0 (0) | 1 (1)
umbilcal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bleeding from hemorrhoids (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 4 (5) | 1 (1)
Difficulty tasting food (General disorders) | 0 (0) | 1 (1)
Edema face (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 4 (7) | 5 (10)
Fatigue (General disorders) | 14 (26) | 15 (28)
Fever (General disorders) | 7 (7) | 3 (5)
Injection site reaction (General disorders) | 2 (2) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (6) | 1 (1)
lightheadedness (General disorders) | 1 (1) | 0 (0)
soft tissue edema (General disorders) | 0 (0) | 1 (1)
hyperbilirubinemia (Hepatobiliary disorders) | 1 (2) | 0 (0)
BK virus (Infections and infestations) | 1 (1) | 0 (0)
C. Diff. infection (Infections and infestations) | 0 (0) | 1 (1)
C. diff. (Infections and infestations) | 0 (0) | 1 (1)
CMV viremia (Infections and infestations) | 1 (2) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
serratia (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lesion on lip after biting lip (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 15 (47) | 10 (18)
Alkaline phosphatase increased (Investigations) | 5 (7) | 4 (13)
Aspartate aminotransferase increased (Investigations) | 13 (34) | 6 (10)
Blood bilirubin increased (Investigations) | 4 (9) | 2 (2)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 14 (25) | 8 (12)
Creatinine increased (Investigations) | 3 (4) | 4 (6)
Lymphocyte count decreased (Investigations) | 20 (81) | 21 (77)
Neutrophil count decreased (Investigations) | 13 (34) | 12 (39)
Platelet count decreased (Investigations) | 19 (78) | 14 (49)
Weight loss (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 18 (63) | 18 (65)
Anorexia (Metabolism and nutrition disorders) | 7 (9) | 6 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 16 (48) | 17 (46)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (3) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 14 (36) | 11 (35)
Hypoalbuminemia (Metabolism and nutrition disorders) | 14 (36) | 7 (18)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (13) | 3 (7)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 12 (37) | 7 (15)
Hypomagnesemia (Metabolism and nutrition disorders) | 16 (46) | 9 (16)
Hyponatremia (Metabolism and nutrition disorders) | 15 (41) | 14 (31)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (8) | 6 (14)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Deconditioning (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (10) | 4 (8)
difficulty dosiflexing rt foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
joint discomfort & instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
shaking chills (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (7) | 4 (8)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 6 (8) | 1 (1)
Lightheadedness (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 4 (7)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (2) | 6 (11)
lightheadedness (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (4) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (7) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (3) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (3) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (3) | 0 (0)
bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Acne Pustules (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (5)
Erythema at injection site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (8)
Pruritis at injection site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (8) | 6 (13)
Purpura (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (5) | 14 (37)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin lesions (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 21 (73) | 19 (74)
Hypotension (Vascular disorders) | 3 (3) | 2 (4)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT02396134/Prot_SAP_000.pdf